CLINICAL TRIAL: NCT00082732
Title: Impact of Dietary Intervention in Men With Hormone Refractory Prostate Cancer
Brief Title: Behavior-Based Dietary Intervention in Treating Patients With Hormone-Refractory Prostate Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000355833; MDA-DM-98054; DM98-054 (Other: UT MD Anderson Cancer Center)
Record Dates: First submitted 2004-05-14; First posted 2004-05-19 (Estimated); Last update posted 2018-11-06 (Actual); Status verified 2018-11

CONDITIONS: Prostate Cancer
Keywords: stage I prostate cancer; stage II prostate cancer; adenocarcinoma of the prostate
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Diet Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm I: Dietary Intervention (Experimental): Nutritional counseling on a low-fat, high-fiber, soy supplemented diet and behavior-based activities, such as goal-setting, contracting, and stimulus control, once weekly for 6 weeks, every 3 weeks for 33 weeks, and then at weeks 44, 48, and 52.
  Interventions: Behavioral: behavioral dietary intervention; Dietary Supplement: dietary intervention; Procedure: therapeutic dietary intervention
- Arm II: Observation (No Intervention): Observation every 6 weeks for 36 weeks and then every 8 weeks for 18 weeks.

INTERVENTIONS:
Behavioral: behavioral dietary intervention
  Arms: Arm I: Dietary Intervention
Dietary Supplement: dietary intervention
  Arms: Arm I: Dietary Intervention
Procedure: therapeutic dietary intervention
  Arms: Arm I: Dietary Intervention

SUMMARY:
RATIONALE: A low-fat, high-fiber diet that includes soy protein may prevent disease progression in patients with hormone-refractory prostate cancer. Nutrition counseling may help motivate patients to follow this diet.

PURPOSE: Randomized phase I trial to study the effectiveness of behavior-based dietary interventions, such as receiving nutrition counseling, in helping patients who have hormone-refractory prostate cancer follow a low-fat, high-fiber, soy-supplemented diet.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine whether a behavior-based dietary intervention can motivate patients with hormone-refractory prostate cancer to adopt and maintain a dietary pattern that includes < 20% of energy from fat, > 25 g of fiber, and 80 g of soy protein powder.
* Compare bioavailable levels of testosterone in patients treated with a behavior-based dietary intervention vs observation only.
* Determine whether this dietary intervention decreases or stabilizes a rising serum prostate-specific antigen level in these patients.
* Determine whether this dietary intervention improves disease-specific survival, mediated by reduced bioavailable levels of testosterone, in these patients.
* Determine the impact of a positive intervention outcome on androgen receptors in patients treated with this dietary intervention.

OUTLINE: This is a randomized, controlled, pilot, multicenter study. Patients are randomized to 1 of 2 treatment arms.

All patients receive nutritional counseling on a healthy diet. Patients also keep a food diary during study participation.

* Arm I (dietary intervention): Patients receive dietary intervention comprising nutritional counseling on a low-fat, high-fiber, soy supplemented diet and behavior-based activities, such as goal-setting, contracting, and stimulus control, once weekly for 6 weeks, every 3 weeks for 33 weeks, and then at weeks 44, 48, and 52. Treatment continues in the absence of disease progression or unacceptable toxicity.
* Arm II (observation): Patients undergo observation every 6 weeks for 36 weeks and then every 8 weeks for 18 weeks.

PROJECTED ACCRUAL: A total of 92 patients (46 per treatment arm) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed adenocarcinoma of the prostate

  * No small cell component
* No histologically confirmed and/or demonstrable metastatic or locally recurrent disease by bone scan, chest x-ray, computed tomography (CT) scan, or transrectal ultrasound

  * No clinical symptoms within the past 90 days
* Documented biochemical failure after radical prostatectomy

  * Prostate-specific antigen must have initially nadired to an undetectable level (< 0.1 ng/mL) after prostatectomy AND is currently rising (0.3-40.0 ng/mL)
* Serum testosterone > 100 ng/dL

PATIENT CHARACTERISTICS:

Age

* Any age

Performance status

* Zubrod 0-1

Life expectancy

* At least 1 year

Hematopoietic

* Not specified

Hepatic

* Not specified

Renal

* Not specified

Other

* No known allergic reactions to milk or soy products

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* More than 1 year since prior chemotherapy

Endocrine therapy

* More than 1 year since prior hormonal therapy

Radiotherapy

* Not specified

Surgery

* See Disease Characteristics

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2000-07-28 (Actual); Primary Completion 2006-02-27 (Actual); Study Completion 2006-02-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard J. Babaian, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas - MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center official website — http://www.mdanderson.org